CLINICAL TRIAL: NCT00685555
Title: SWITCH: Rationale, Design, and Implementation of a Community, School, and Family-based Intervention to Modify Behaviors Related to Childhood Obesity
Brief Title: Healthy Futures Project: A Community Based Obesity Prevention Program
Acronym: SWITCH
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Media and the Family (Other)
Collaborators: Fairview Health Services (Other); Medica (Unknown); Healthy and Active America Foundation, (Unknown); Cargill (Industry); Spunk Design Machine (Unknown); Iowa State University (Other); Michigan State University (Other); University of Minnesota (Other)
Responsible Party: Dr. David Walsh, President and Founder, National Institute on Media and the Family
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIMF-1300-05
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2008-05

CONDITIONS: Overweight; Obesity
Keywords: Screen time; Fruits and Vegetable Consumption; Physical Activity; Obesity; Overweight
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Switch active lifestyles brought to you by MediaWise — The Switch™ Program is a unique community and family-based behavior change initiative that helps motivate children to change three critical health behaviors that are risk factors for childhood overweight and obesity.
  Other Names: Iowa State University; Michigan State University; National Institute on Media and the Family
Behavioral: Switch active lifestyles from MediaWise — 1300 students (male and female) were recruited through two separate school districts in Lakeville, Minnesota and Cedar Rapids, Iowa. Informed consents went to all students who chose to participate. Demonstration and Control school were randomly selected. Baseline data was collected regarding physical activity, screen time, and nutrition, standard body measurements, and baseline data, and salivary cortisol levels were taken. Parent and teacher surveys were also conducted. After baseline selected demonstration sites and students were provided with information focused on improving healthy behaviors while the control sites served as matched comparison groups.
  Other Names: Switch; Switch program; The Switch program

SUMMARY:
The purpose of this research is to increase community awareness about the relationship between physical activity, screen time, and nutrition and how these factors influence healthy weight management.

The problem of obesity is at epidemic proportions and has become the most important public health problem confronting the United States today. Of greatest concern is the 300% increase in obesity rates among children and youth over the past twenty years. Childhood obesity is a precursor of adult obesity.

DETAILED DESCRIPTION:
The Switch™ Program is a unique community and family-based behavior change initiative that helps motivate children to change three critical health behaviors that are risk factors for childhood overweight and obesity. Through community education, family-based strategies and partnerships with schools, 3rd, 4th and 5th graders are encouraged to: Switch what you Do™ Switch what you View™ Switch what you Chew™.

ELIGIBILITY:
Inclusion Criteria:

* All children in 3-5 grades who provide parental consent and child assent will be eligible to participate in the project.

Exclusion Criteria:

* Participants who meet the following exclusion criteria will not be considered for participation.
* Do not provide consent
* unable or unwilling to adhere to project procedures

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1300 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Our outcome measure was reduction of screen time | 4 waves of data

SECONDARY OUTCOMES:
Our secondary outcome measure increase in fruit and vegetable consumption. | T1-PRE Intervention toT2 Post Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dave Walsh, Ph.D., Principal Investigator — National Institute on Media and the Family
Locations (1):
- National Institute on Media and the Family, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Eisenmann JC, Laurson KR, Wickel EE, Gentile D, Walsh D. Utility of pedometer step recommendations for predicting overweight in children. Int J Obes (Lond). 2007 Jul;31(7):1179-82. doi: 10.1038/sj.ijo.0803553. Epub 2007 Jan 30. PMID 17264846
- [Derived] Eisenmann JC, Gentile DA, Welk GJ, Callahan R, Strickland S, Walsh M, Walsh DA. SWITCH: rationale, design, and implementation of a community, school, and family-based intervention to modify behaviors related to childhood obesity. BMC Public Health. 2008 Jun 29;8:223. doi: 10.1186/1471-2458-8-223. PMID 18588706
- See also: National Institute on Media and the Family — http://www.mediawise.org
- See also: Co-Investigator Douglas Gentile Ph.D. — http://www.psychology.iastate.edu/index.php?id=61